CLINICAL TRIAL: NCT03219918
Title: Adenoma Detection Rate in Colonoscopy Performed With EndoRings - a Single-centre Prospective Randomised Clinical Trial
Brief Title: Adenoma Detection Rate in Colonoscopy Performed With EndoRings
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Practically difficult to inroll the number of patients anticipated
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ZUH-KØGE-KIR1
Record Dates: First submitted 2017-06-13; First posted 2017-07-18 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Colorectal Adenoma; Colorectal Neoplasms
Keywords: Colorectal adenoma; Colonoscopy; Caps; Adenoma detection rate
MeSH Terms: conditions — Colorectal Neoplasms; Cryopyrin-Associated Periodic Syndromes

STUDY DESIGN:
Intervention Model Description: The study is a single-centre prospective randomised clinical trial. Patients are included if they meet the specified inclusion criteria and accept to take part in the study after proper oral and written information (see patient information below).
  Specimens i.e. removed adenomas and biopsies of suspected malignancies are analysed by pathologists according to standard procedure. The pathologist will not know the nature of specimen collection (colonoscopy with or without EndoRings). The specimens are not saved for any other study related activities.
Who Masked: Investigator, Outcomes Assessor
Masking Description: It is partially blinded in the way that the endoscopist knows whether the procedure is performed with or without the EndoRings but neither patient, pathologist nor investigators will have this information, which is only to be revealed to the investigators at the end of data processing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With EndoRings (Active Comparator): Colonoscopy is performed with the use of the cap-device EndoRings II Distal Attachment to be attached to the tip of the colonoscope
  Interventions: Device: EndoRings II Distal Attachment
- NO EndoRings (No Intervention): Colonoscopy is performed conventionally without any caps

INTERVENTIONS:
Device: EndoRings II Distal Attachment — Colonoscopy cap
  Arms: With EndoRings

SUMMARY:
The study is designed to examine whether colonoscopy using an EndoRings cap has a higher adenoma detection rate than conventional colonoscopy. Secondary end-points is to compare completion rate, completion time, complication rate and detection of malignancies. Half of the patients will be randomised to colonoscopy using cap and the other half to no cap.

DETAILED DESCRIPTION:
Colonoscopy is recognised as the standard method for finding and removing colorectal adenomas, which are precursors of most colorectal cancers. It has been shown that there is a direct correlation between adenoma detection rate and the risk of developing colorectal cancer subsequently. However, patients undergoing colonoscopy are still at risk of developing colorectal cancer, mainly because precursor lesions are missed during the procedure. This may be due to insufficient bowel preparation, difficulties in visualising flat lesions or the location of lesions behind haustral folds.

Improving the ADR can be achieved by different means; better training of endoscopists, improved bowel preparation, optimal sedation and medico technical developments. The technical improvements have mainly been in the optimising of image and improved scope thickness and flexibility, including devices that improve visualisation by increasing the exposed colonic surface . One of these new inventions is the EndoRings II Distal Attachment.

According to the Danish Colorectal Cancer Screening Database, the ADR of standard screening colonoscopy is between 34 and 67 % with a national average of 49 % of patients with detected adenomas. Due to the known adenoma miss rate in standard screening colonoscopies, it is important to increase the ADR on average as well as finding ways to improve ADR for centres with a lower than average ADR.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all the below listed criteria are eligible for inclusion in the trial:

1. Age between 50 - 74 years (age range of screening population)
2. Positive HemoCult home test from the Danish Colorectal Cancer Screening Programme
3. Ability to give informed consent to participation in the trial.

Exclusion Criteria:

Patients meeting one or more of the below listed criteria will be excluded from the trial:

1. History of colorectal cancer
2. History of Inflammatory Bowel Disease
3. Part of other control programme (e.g. HNPCC or adenoma control)
4. ASA =/> 4 and/or necessity of general anaesthesia
5. Former surgery with removal of a part of the colon on either benign or malignant background

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | maximum 60 minutes
  Number of colorectal adenomas/neoplasms/carcinomas found in colonoscopy

SECONDARY OUTCOMES:
Completion time | maximum 60 minutes
  Overall colonoscopy duration
Completion rate | maximum 60 minutes
  Colonoscopy completion (intubation to coecum)
Malignancy detection | maximum 60 minutes
  Number of colorectal malignancies found in colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Line E Line, MD, Principal Investigator — Zealand University Hospital Køge; Ismayil Gögenur, Prof, DMSc, Study Director — Zealand University Hospital Køge
Locations (1):
- Zealand University Hospital Køge, Department of Surgery, Køge, Denmark

IPD SHARING:
Plan to Share IPD: Undecided